CLINICAL TRIAL: NCT01680497
Title: Post-Market Study of JUVÉDERM VOLIFT™ With Lidocaine for the Correction of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAF/AGN/MED/FIL/018
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Moderate to Severe Nasolabial Folds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JUVÉDERM VOLIFT™ (Experimental): All subjects receiving treatment with JUVÉDERM VOLIFT™.
  Interventions: Device: Crosslinked hyaluronic acid dermal filler

INTERVENTIONS:
Device: Crosslinked hyaluronic acid dermal filler — All treatment details are at the discretion of the Investigator and should be guided by the Directions for Use. Up to 3 treatments will be administered: Initial treatment, optional top-up treatment at Day 14 post-initial treatment, and optional repeat treatment at Month 12 post-initial treatment.
  Other Names: JUVÉDERM VOLIFT™

SUMMARY:
A prospective, open-label, multi-center, observational, post-market study evaluating JUVÉDERM VOLIFT™ for the correction of moderate to severe nasolabial folds

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Have 2 fully visible, approximately symmetrical nasolabial folds and has severity scores of 2 or 3 on the 5-point photographic nasolabial fold severity scale (range 0-4) for both nasolabial folds, as judged by the Investigator
* Have a reasonable expectation for correction by injection via deep dermis, as described in the protocol
* Agree to refrain from undergoing other anti-wrinkle/volumizing treatments in the lower two-thirds of the face (below the orbital rim) for the duration of the study
* Understand and be willing to follow all aspects of the study protocol and have signed and dated the Informed Consent prior to any study-related procedures being performed
* Be in good health as in the opinion of the Investigator

Exclusion Criteria:

* Has undergone cosmetic facial procedures (e.g., face lift or other surgeries) which may alter the appearance of the nasolabial fold area
* Cosmetic injections in the lower two-thirds of the face (below the orbital rim), within 6 months prior to entry in the study, or be planning to undergo any of these procedures at any time during the study. NOTE: Prior treatment with HA fillers and/or collagen is allowed, provided the treatment was administered more than 6 months prior to study entry
* Has undergone volumizing of the mid/lower face within 9 months prior to study entry
* Has ever received semi-permanent fillers or permanent facial implants (e.g., calcium hydroxylapatite, poly-L-lactic acid, polymethylmethacrylate, silicone, expanded poly-tetrafluoroethylene) anywhere in the lower face (below the orbital rim), or be planning to be implanted with any of these products at any time during the study
* Have a history of anaphylaxis, multiple severe allergies, atopy, allergy to lidocaine (an any amide-based anesthetics), HA products, or Streptococcal protein, or be planning to undergo a desensitization therapy during the term of the study
* Be a pregnant female, lactating, or planning to become pregnant at any time during the study
* Be a female of childbearing potential not using a reliable means of contraception
* Have received any investigational product within 30 days prior to study enrollment or be planning to participate in another investigation during the course of this study
* Suffer from an uncontrolled personality disorder (e.g., body dysmorphia, depression)
* Have a history of or currently suffer from autoimmune disease (e.g., rheumatoid arthritis, Crohn's disease)
* Have a history of streptococcal disease (e.g., strep throat or rheumatic fever with or without heart complications)
* Have a history of skin cancer
* Suffer from porphyria
* Have epilepsy, which is not controlled by anti-epilepsy therapy
* Current cutaneous inflammatory and/or infectious processes (e.g., acne, herpes)
* Have a history of treatment with interferon
* Be on an ongoing regimen of anti-coagulation therapy (e.g., warfarin) or have taken non-steroidal anti-inflammatory drugs (NSAIDs) (e.g., aspirin, ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with garlic or ginkgo biloba) within 10 days of undergoing study device injection. NOTE: Study device injection may be delayed as necessary to accommodate this 10-day period
* Be on a concurrent regimen of high doses of lidocaine (more than 400 mg) which may cause acute toxic reactions
* Be on a concurrent regimen of other local anesthetics structurally related to amide-type local anesthetics
* Have impaired cardiac conduction, severely impaired hepatic function, or severe renal dysfunction
* Have a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2014-03-06 (Actual); Study Completion 2014-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Allergan Medical
Locations (3):
- Germany (2):
  - Cologne
  - Darmstadt
- Naarden, Netherlands

REFERENCES:
- [Background] Sattler G, Philipp-Dormston WG, Van Den Elzen H, Van Der Walt C, Nathan M, Kolodziejczyk J, Kerson G, Dhillon B. A Prospective, Open-Label, Observational, Postmarket Study Evaluating VYC-17.5L for the Correction of Moderate to Severe Nasolabial Folds Over 12 Months. Dermatol Surg. 2017 Feb;43(2):238-245. doi: 10.1097/DSS.0000000000000939. PMID 28165349

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | JUVÉDERM VOLIFT™
Started | 70
Completed | 68
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | JUVÉDERM VOLIFT™
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Investigator Assessment of Nasolabial Fold Severity Using the 5-point Nasolabial Fold Severity Scale (NLFSS)
Description: Nasolabial fold severity is evaluated by the Investigator on the 5-point NLFSS on both the right and left sides. Scores are assessed as 1 (none), 2 (mild), 3 (moderate), 4 (severe), and 5 (extreme).
Time Frame: Month 12
Population: Efficacy Population: all subjects who completed their first treatment session as planned, had no major protocol violations that would potentially affect outcome measures, and had data at the time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | JUVÉDERM VOLIFT™
Number analyzed (Participants) | 65
Scores on a Scale
  12 Months - Right | 2.8 (0.8)
  12 Months - Left | 2.8 (0.8)

2. Secondary Outcome: Investigator Assessment of Nasolabial Fold Severity Using the 5-point NLFSS
Description: as for outcome 1
Time Frame: Day 0, Day 14, Month 1, Month 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | JUVÉDERM VOLIFT™
Number analyzed (Participants) | 67
Scores on a Scale
  Day 0 - Right | 3.6 (0.5)
  Day 0 -Left | 3.7 (0.5)
  Day 14 - Right | 1.7 (0.5)
  Day 14 - Left | 1.7 (0.5)
  Month 1 - Right (N=66) | 1.8 (0.6)
  Month 1 - Left (N=66 | 1.9 (0.6)
  Month 9 - Right (N=66) | 2.5 (0.7)
  Month 9 - Left (N=66) | 2.4 (0.7)

3. Secondary Outcome: Investigator Satisfaction With Aesthetic Outcome on an 11-Point Scale
Description: Investigator satisfaction with aesthetic outcome is assessed on an 11-point scale. Scores range from -5 (definitely not satisfied), 0 (don't know/unsure), and 5 (definitely satisfied).
Time Frame: Day 14, Month 1, Month 9, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | JUVÉDERM VOLIFT™
Number analyzed (Participants) | 67
Scores on a Scale
  Day 14 | 4.6 (0.6)
  Month 1 (N=66) | 4.5 (0.7)
  Month 9 (N=65) | 4.0 (1.1)
  Month 12 (N=65) | 4.4 (1.0)

4. Secondary Outcome: Investigator Assessment of Ease of Injection Use on a 10-Point Scale
Description: Investigator assessment of ease of injection use is assessed on a 10-point scale. Scores range from 0 (easy) to 10 (hard).
Time Frame: Day 0, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | JUVÉDERM VOLIFT™
Number analyzed (Participants) | 67
Scores on a Scale
  Day 0 | 1.2 (1.3)
  Day 14 (N=27) | 0.9 (0.5)

5. Secondary Outcome: Subject Assessment of Nasolabial Fold Severity Using the 5-point NLFSS
Description: Nasolabial fold severity is evaluated by the subject on the 5-point NLFSS on both the right and left sides. Scores are assessed as 1 (none), 2 (mild), 3 (moderate), 4 (severe), and 5 (extreme).
Time Frame: Day 0, Day 14, Month 1, Month 9, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | JUVÉDERM VOLIFT™
Number analyzed (Participants) | 67
Scores on a Scale
  Day 0 - Right | 3.8 (0.7)
  Day 0 - Left | 3.9 (0.7)
  Day 14 - Right | 1.8 (0.7)
  Day 14 - Left | 1.8 (0.7)
  Month 1 - Right (N=66) | 2.0 (0.9)
  Month 1 - Left (N=65) | 2.1 (0.8)
  Month 9 - Right (N=66) | 2.6 (0.8)
  Month 9 - Left (N=66) | 2.6 (0.8)
  Month 12 - Right (N=54) | 2.9 (0.8)
  Month 12 - Left (N=54) | 3.0 (0.9)

6. Secondary Outcome: Subject Satisfaction With Aesthetic Outcome on an 11-Point Scale
Description: Subject satisfaction with aesthetic outcome is assessed on an 11-point scale. Scores range from -5 (definitely not satisfied), 0 (don't know/unsure), and 5 (definitely satisfied).
Time Frame: Day 14, Month 1, Month 9, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | JUVÉDERM VOLIFT™
Number analyzed (Participants) | 67
Scores on a Scale
  Day 14 | 4.2 (1.0)
  Month 1 (N=66) | 4.2 (1.0)
  Month 9 (N=66) | 3.2 (2.4)
  Month 12 (N=54) | 3.3 (1.9)

7. Secondary Outcome: Subject Assessments of Pain, Swelling, and Bruising Intensity on an 11-Point Scale
Description: Subject assessment of pain, swelling and bruising intensity on an 11-point scale. Scores range from 0 (No pain/swelling/bruising) to 10 (worst pain/swelling/bruising imaginable).
Time Frame: Day 0, Day 14, Month 12, Month 12.5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | JUVÉDERM VOLIFT™
Number analyzed (Participants) | 67
Scores on a Scale
  Pain Intensity Day 0 - Right | 2.0 (1.8)
  Pain Intensity Day 0 - Left | 2.0 (1.8)
  Pain Intensity Day 14 - Right (N=66) | 0.8 (1.7)
  Pain Intensity Day 14 - Left (N=66) | 0.7 (1.5)
  Pain Intensity Month 12 - Right (N=51) | 1.5 (1.8)
  Pain Intensity Month 12 - Left (N=51) | 1.5 (2.1)
  Pain Intensity Month 12.5 - Right (N=12) | 0.0 (0.0)
  Pain Intensity Month 12.5 - Left (N=12) | 0.0 (0.0)
  Swelling Intensity Day 0 - Right | 1.7 (1.6)
  Swelling Intensity Day 0 - Left | 1.7 (1.6)
  Swelling Intensity Day 14 - Right (N=66) | 1.5 (2.2)
  Swelling Intensity Day 14 - Left (N=66) | 1.4 (2.2)
  Swelling Intensity Month 12 - Right (N=51) | 1.4 (1.5)
  Swelling Intensity Month 12 - Left (N=51) | 1.4 (1.6)
  Swelling Intensity Month 12.5 - Right (N=12) | 0.1 (0.3)
  Swelling Intensity Month 12.5 - Left (N=12) | 0.2 (0.4)
  Bruising Intensity Day 0 - Right | 0.3 (0.9)
  Bruising Intensity Day 0 - Left | 0.3 (0.9)
  Bruising Intensity Day 14 - Right (N=66) | 0.9 (1.9)
  Bruising Intensity Day 14 - Left (N=66) | 0.5 (1.3)
  Bruising Intensity Month 12 - Right (N=51) | 0.4 (0.8)
  Bruising Intensity Month 12 - Left (N=51) | 0.4 (0.9)
  Bruising Intensity Month 12.5 - Right (N=12) | 0.3 (0.7)
  Bruising Intensity Month 12.5 - Left (N=12) | 0.5 (0.8)

ADVERSE EVENTS:
Description: The Safety Population is used to assess adverse events (AEs) and serious adverse events (SAEs) and includes all treated subjects.
Arm/Group | JUVÉDERM VOLIFT™
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.